CLINICAL TRIAL: NCT02597881
Title: Registry of Patients With Bone Disorders
Brief Title: Achondroplasia Natural History Multicenter Clinical Study
Status: Suspended | Type: Observational
Why Stopped: Did not renew protocol before expiration date. PI error. Currently communicating with local IRB as to process to reinstate protocol or create new, replacement protocol.
Sponsor: Johns Hopkins University (Other)
Collaborators: University of Wisconsin, Madison (Other); Alfred I. duPont Hospital for Children (Other); University of Texas (Other); BioMarin Pharmaceutical (Industry); Greenberg Center for Skeletal Dysplasias (Unknown)
Responsible Party: Sponsor
Other Study IDs: NA_00086185
Record Dates: First submitted 2015-10-26; First posted 2015-11-05 (Estimated); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Achondroplasia
Keywords: natural history
MeSH Terms: conditions — Achondroplasia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to create an electronic registry to house phenotypic information from patients with achondroplasia. The initial focus of this registry will be to include U.S. patients with achondroplasia. Once populated, the collective data can be queried to pursue clinical research questions pertaining to health outcomes and treatment options for patients with this conditions. The registry is longitudinal in nature with the functionality to retrospectively enter patients' clinical data from the prenatal period up through the most recent encounter, with all intervening data entered in a chronologic fashion.

DETAILED DESCRIPTION:
The purpose of this protocol is to create an electronic registry to house phenotypic information from patients with all types of bone conditions. The initial focus of this registry will be to include U.S. patients with achondroplasia. Once populated by co-investigators with particular interest, expertise and large clinical populations with these bone conditions, the collective data can be queried to pursue clinical research questions pertaining to health outcomes and treatment options for patients with these complex conditions. The registry is longitudinal in nature with the functionality to retrospectively enter patients' clinical data from the prenatal period up through the most recent encounter, with all intervening data entered in a chronologic fashion. The database has been created in RedCap, a publicly available database format created by researchers at the University of Miami specifically for academic researchers collaborating across multiple research sites. The rationale for creating such a database is simple; achondroplasia is relatively rare so collaboration among researchers is essential to gather similarly affected patients to answer common clinical research questions. The goal is to better understand the natural history and treatment outcomes for these patients.

This registry was built by, based at and maintained by personnel from the Greenberg Center for Skeletal Dysplasias in the McKusick-Nathans Institute of Genetic Medicine (IGM) at Johns Hopkins. The registry is web-based and therefore easily accessible to our co-investigators at other sites across the U.S., including Alfred I. DuPont in Wilmington, Delaware, University of Wisconsin in Madison and University of Texas.

Our goal is to enroll at least 1500 patients with achondroplasia from the aforementioned sites. Access to the registry is password-protected and the data will be backed up on the IGM server daily. A co-investigator will be able to enter and access the identifying information (i.e. name, address, contact information, DOB) for their patients only in the registry. Thereafter, a unique study identification number, calculated age of the subject (based on the date of data entry) and diagnosis will be the only identifiers accessible to the other co-investigators. The total deidentified phenotype data will be available to the co-investigators during data analysis.

ELIGIBILITY:
Inclusion Criteria:

* Molecular or clinical diagnosis of achondroplasia (as confirmed by physical exam and/or radiograph review by the PI, one of the co-PIs or other qualified clinical geneticists)
* Subjects must have been seen for a clinical genetics visit at Johns Hopkins, Alfred I. DuPont Hospital for Children, University of Wisconsin-Madison or University of Texas
* Subjects may be active clinical patients at the above sites or no longer treated at a given site but with sufficient retrospective clinical data for extraction as determined by the PI or co-PIs

Exclusion Criteria:

* Skeletal dysplasia diagnosis other than heterozygous
* Achondroplasia
* There is no medical complication or condition which excludes a patient with achondroplasia

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Achondroplasia patients seen at one of the participating sites
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2016-04 (Actual); Primary Completion 2024-12 (Actual); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Collection of growth measurements of patients with Achondroplasia using chart reviews | 3 years
  Determine age at which linear growth ceases in patients with achondroplasia by gender

SECONDARY OUTCOMES:
Number of surgeries undertaken by achondroplasia patients using chart reviews. | 3 years
  To quantify the total number, type, age indications and complications of all surgical interventions of a cohort of patients with achondroplasia

CONTACTS AND LOCATIONS:
Overall Officials: Julie Hoover-Fong, MD,PhD, Principal Investigator — Johns Hopkins University

IPD SHARING:
Plan to Share IPD: No